CLINICAL TRIAL: NCT00094601
Title: Cognitive Function in Parkinson's Disease: Relationship to Cortical Dopamine Synthesis and Dopamine D1 Receptors
Brief Title: Relationship of Dopamine to Cognitive Function in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050011; 05-M-0011
Record Dates: First submitted 2004-10-20; First posted 2004-10-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-01-22

CONDITIONS: Parkinson Disease
Keywords: Positron Emission Tomograhy; [18F] FDOPA; [11C] NNC-112; Dopamine; Molecular Imaging; Dopamine D1 Receptor; PET; Parkinson's Disease; Cognition; Parkinson Disease; PD; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
This study will examine how the brain chemical dopamine affects memory, reasoning, and other thought processes in people with Parkinson's disease with and without dementia and in healthy control subjects.

Healthy normal volunteers and people with Parkinson's disease who are between 40 and 85 years of age may be eligible for this study. Pregnant women with Parkinson's disease and breastfeeding normal volunteers are excluded. Candidates are screened with a physical and neurological examination, blood tests, a brief mental test called the Mini Mental Status Examination, and other tests designed to assess memory, learning, reasoning, and other thought processes. Patients with Parkinson's disease also undergo a more thorough mental evaluation called the Mattis Dementia Rating Scale. The study requires about 15 hours over 4 or 5 outpatient visits to NIH.

Participants undergo two positron emission tomography (PET) scans on two separate days and a magnetic resonance imaging (MRI) scan, as follows:

PET Scans

The two PET procedures are done the same way, except one uses a radioactive tracer called [(18)F]DOPA and one uses a tracer called [(11)C]NNC-112. A catheter (small plastic tube) is placed in a vein in the subject's arm for injection of the tracer. The subject lies on the scanner bed and a special mask is fitted to his or her head to hold it in place during the procedure. Just before injecting the tracer, a 10-minute "transmission scan" is done of the head using a tracer called (68)Ge. Then, a series of scans using one of the two study tracers ([(18)F]DOPA or [(11)C]NNC-112 are done for about 90 minutes. About 1 hour before injection of the [(18)F]DOPA tracer, subjects take 200 mg of the drug carbidopa by mouth to help the tracer work properly. Blood pressure, breathing and heart are monitored before and after injection of the [(11)C]NNC-112 tracer.

Patients with Parkinson's disease are taken off all Parkinson's medications the night before the [(18)F]DOPA scan and their motor function is tested the following morning before the scans are done, using the Unified Parkinson's Disease Rating Scale. Patients can resume all medications except L-DOPA (including Sinemet) after the movement test, and they can resume L-DOPA after the PET scan is finished.

MRI Scan

MRI uses a strong magnetic field and radio waves to obtain images of the brain. The subject lies still on a table that slides inside the scanner, a metal cylinder. They wear ear plugs to muffle loud knocking sounds that occur during the scanning and can communicate with the MRI staff at any time through an intercom.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disorder, particularly in the elderly population. PD is characterized primarily by motor impairment, but cognitive impairment is common and dementia may occur in about 30% of patients. The pathological hallmark of PD is the selective degeneration of nigrostriatal dopamine neurons and the appearance of intracytoplasmic inclusions known as Lewy Bodies. Dopaminergic dysfunction has been widely demonstrated in PD patients. Reductions in [18F]FDOPA uptake has been consistently observed in PD, although it remains to be established whether there are relative differences between PD with and without dementia, and its association with cognitive function. Furthermore, data relating to dopamine D1 receptors in PD are limited to post mortem studies and imaging with the D1 tracer [11C]SCH 23390, and little is known about the role of D1 receptors in vivo and how it relates to clinical phenomena. The aim of the current study is to assess the feasibility and usefulness of imaging of the dopamine D1 receptor and dopamine terminal function in vivo, using PET (positron emission tomography) in patients with PD, with and without dementia, and to assess changes in presynaptic and postsynaptic dopaminergic markers in PD. The long-term goal of the present study is to further our understanding of the role of the dopaminergic system in the pathogenesis of PD and its relationship with cognitive and motor deficits of PD. Knowledge gained from the present study may assist in the development of novel therapeutic targets for PD.

ELIGIBILITY:
* INCLUSION CRITERIA:

PD patients must meet the diagnosis of idiopathic Parkinson's disease. Diagnosis will be based upon the presence of at least two of the four cardinal symptoms (tremor, bradykinesia, rigidity and instability) as well as a positive response to dopaminergic agents.

Patients will be on stable dopaminergic therapy for approximately two weeks prior to enrollment.

Control subjects must be healthy and aged 40 - 85 years and will be age and gender matched to PD patients.

EXCLUSION CRITERIA - CONTROLS:

Diagnosis of idiopathic Parkinson's disease.

Secondary cause of Parkinsonism, e.g. Wilson's disease, neuroleptic use.

Psychiatric disease that would, in judgment of the investigator, interfere with the safe conduct of the study.

Current psychiatric illness.

Severe depressive symptoms with BDI 16+.

Substance abuse, severe systemic disease, poor vision or hearing based on history and physical exam.

Incidence of Parkinson's disease in two or more first degree relatives.

Dementia not due to PD or severe dementia with MMSE less than 15.

Neurological disorder other than PD that would effect protocol (e.g. stroke, Alzheimer's disease).

Laboratory tests with clinically significant abnormalities.

History of an abnormal MRI.

Pregnancy or breast feeding.

Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual NIH RSC limits.

Any conditions that increase risk for MRI (pacemaker, metallic foreign body, claustrophobia, etc.).

Any medical condition that in the opinion of the investigators would interfere with the safe conduct of the study.

Severe hypertension. The subject may be on anti-hypertensive medications. The initial screening must show no more than moderate hypertension - i.e. less than 160/95. In addition, the subject must have normal laboratory values (e.g., BUN, creatinine, urinalysis, and ECG) to document lack of end organ damage. On baseline evaluation on the day of the scan (i.e., before injection of tracer), the subject must be asymptomatic (no headache, dizziness, neurological symptoms, or blurred vision) AND have sustained BP less than 180/100.

Inability to provide consent.

Smoking within 6 months prior to enrollment in the study.

EXCLUSION CRITERIA - PATIENTS:

Secondary cause of Parkinsonism, e.g. Wilson's disease, neuroleptic use.

Psychiatric disease that would, in judgment of the investigator, interfere with the safe conduct of the study.

Current psychiatric illness except for depression.

Severe depressive symptoms with BDI 16+.

Substance abuse, severe systemic disease, poor vision or hearing based on history and physical exam.

Dementia not due to PD or severe dementia with MMSE less than 15.

Neurological disorder other than PD that would effect protocol (e.g. stroke, Alzheimer's disease).

Laboratory tests with clinically significant abnormalities.

History of an abnormal MRI.

Pregnancy or breast feeding.

Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual NIH RSC limits.

Any conditions that increase risk for MRI (pacemaker, metallic foreign body, claustrophobia, etc.).

Any medical condition that in the opinion of the investigators would interfere with the safe conduct of the study.

Severe hypertension. The subject may be on anti-hypertensive medications. The initial screening must show no more than moderate hypertension - i.e. less than 160/95. In addition, the subject must have normal laboratory values (e.g., BUN, creatinine, urinalysis, and ECG) to document lack of end organ damage. On baseline evaluation on the day of the scan (i.e., before injection of tracer), the subject must be asymptomatic (no headache, dizziness, neurological symptoms, or blurred vision) AND have sustained BP less than 180/100.

Inability to provide consent.

Smoking within 6 months prior to enrollment in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2004-10-18; Study Completion 2008-01-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Mawlawi O, Lombardo I, Gil R, Martinez D, Huang Y, Hwang DR, Keilp J, Kochan L, Van Heertum R, Gorman JM, Laruelle M. Prefrontal dopamine D1 receptors and working memory in schizophrenia. J Neurosci. 2002 May 1;22(9):3708-19. doi: 10.1523/JNEUROSCI.22-09-03708.2002. PMID 11978847